CLINICAL TRIAL: NCT05564130
Title: Bicarbonate for In-Hospital Cardiac Arrest - A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Bicarbonate for In-Hospital Cardiac Arrest
Acronym: BIHCA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lars Wiuff Andersen (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Lars Wiuff Andersen, Associate Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00004
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium bicarbonate (Experimental): 50 ml of 1 mmol/ml sodium bicarbonate given as soon as possible after the first dose of adrenaline. If the patient remains in cardiac arrest, one additional dose of 50 ml of 1 mmol/ml sodium bicarbonate will be administered after the second dose of adrenaline dose for a maximum of two doses.
  Interventions: Drug: Sodium bicarbonate
- Placebo (Placebo Comparator): 50 mL of 9 mg/mL NaCl ("normal saline") given as soon as possible after the first dose of adrenaline. If the patient remains in cardiac arrest, one additional dose of 50 mL of 9 mg/mL NaCl will be administered after the second dose of adrenaline dose for a maximum of two doses.
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Sodium bicarbonate — Sodium bicarbonate 1 mmol/ml
  Arms: Sodium bicarbonate
Drug: Sodium chloride — Sodium chloride 9 mg/mL
  Arms: Placebo

SUMMARY:
This is an investigator-initiated, multicenter, randomized, placebo-controlled, parallel group, double-blind, superiority trial of sodium bicarbonate during adult in-hospital cardiac arrest. There will be 22 enrolling sites in Denmark. 778 adult patients with in-hospital cardiac arrest receiving at least one dose of adrenaline will be enrolled. The primary outcome is return of spontaneous circulation and key secondary outcomes include survival at 30 days and survival at 30 days with a favorable neurological outcome.

ELIGIBILITY:
Inclusion Criteria:

1. In-hospital cardiac arrest
2. Age ≥ 18 years
3. Received at least one dose of adrenaline during cardiopulmonary resuscitation (CPR)

Exclusion Criteria:

1. Clearly documented "do-not-resuscitate" order prior to the cardiac arrest
2. Prior enrollment in the trial
3. Invasive mechanical circulatory support at the time of the cardiac arrest
4. Known or suspected pregnancy at the time of the cardiac arrest
5. Known objection by the patient to participate in the trial
6. Clinical indication for bicarbonate administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 778 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-05-28 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Return of Spontaneous Circulation | During the cardiac arrest, an average of 20 minutes
  Return of spontaneous circulation is defined as spontaneous circulation with no further need for chest compressions sustained for at least 20 minutes

SECONDARY OUTCOMES:
Number of Participants That Survived 30 Days | At 30 days
Number of Participants With a Favorable Neurological Outcome at 30 Days | At 30 days
  A favorable neurological outcome will be defined as a modified Rankin Scale score of 0, 1, 2 or 3. The modified Rankin Scale is a 7-point scale assessing neurological/functional outcomes after brain damage with higher scores indicating worse neurological/functional outcomes.

OTHER OUTCOMES:
Survival | At 90 days, 180 days, and 1 year
Favorable Neurological Outcome | At 90 days, 180 days, and 1 year
  A favorable neurological outcome will be defined as a modified Rankin Scale score of 0, 1, 2 or 3. The modified Rankin Scale is a 7-point scale assessing neurological/functional outcomes after brain damage with higher scores indicating worse neurological/functional outcomes.
Health-related Quality of Life (EQ-5D-5L) | At 30 days, 90 days, 180 days, and 1 year
  The EQ-5D-5L is a well-established measure of health-related quality of life that is quantified as a utility (i.e. a measure of quality of life between 0 and 1).
Cerebral performance category | At 30 days, 90 days, 180 days, and 1 year
  The cerebral performance category score is a 5-point scale assessing neurological/functional outcomes after brain damage with higher scores indicating worse neurological/functional outcomes.
Sequential Organ Failure Assessment (SOFA) Score | At 2, 24, 48 and 72 hours
  The SOFA score is a validated and widely used measure of organ failure assessing the respiratory, nervous, cardiovascular, hepatic, coagulation, and renal systems. We will assess both the cardiovascular sub score as well as the overall SOFA score.
Hospital Disposition | At hospital discharge, up to 1 year
  Hospital disposition (e.g. home, rehabilitation, nursing home, hospice) will be defined at the time of discharge from the initial acute care hospital.
pH | Immediately after return of spontaneous circulation, often within 1 hour
  Unit: None
Standard bicarbonate | Immediately after return of spontaneous circulation, often within 1 hour
  Unit: mmol/L
pCO2 | Immediately after return of spontaneous circulation, often within 1 hour
  Partial pressure of CO2 in arterial blood. Unit: kPa
Potassium | Immediately after return of spontaneous circulation, often within 1 hour
  Unit: mmol/L
Calcium | Immediately after return of spontaneous circulation, often within 1 hour
  Unit: mmol/L
Sodium | Immediately after return of spontaneous circulation, often within 1 hour
  Unit: mmol/L
Lactate | Immediately after return of spontaneous circulation, often within 1 hour
  Unit: mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Lars W Andersen, Principal Investigator — Aarhus University Hospital
Locations (22):
- Denmark (22):
  - Hospital of Southern Jutland - Aabenraa, Aabenraa
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Copenhagen University Hospital - Bispebjerg, Bispebjerg
  - Copenhagen University Hospital - Rigshospitalet, Copenhagen
  - Hospital of Southwest Jutland - Esbjerg, Esbjerg
  - Copenhagen University Hospital - Gentofte, Gentofte Municipality
  - Gødstrup Hospital, Gødstrup
  - Copenhagen University Hospital - Herlev, Herlev
  - North Denmark Region Hospital - Hjørring, Hjørring
  - Holbæk Hospital, Holbæk
  - Horsens Regional Hospital, Horsens
  - Hvidovre Hospital, Hvidovre
  - Kolding Hospital, Kolding
  - Zealand University Hospital - Køge, Køge
  - Nykøbing Falster Hospital, Nykøbing Falster
  - Odense University Hospital, Odense
  - Randers Regional Hospital, Randers
  - Zealand University Hospital - Roskilde, Roskilde
  - Slagelse Hospital, Slagelse
  - Odense University Hospital - Svendborg, Svendborg
  - Viborg Regional Hospital, Viborg

IPD SHARING:
Plan to Share IPD: Yes
Six months after the publication of the last results, all de-identified individual patient data will be made available for data sharing. Procedures, including re-coding of key variables, will be put in place to allow for complete de-identification of the data. Data will be completely anonymized according to Danish law.
  All relevant trial-related documents, including the protocol, data dictionary, and the main statistical code, will be shared along with the data. There will be no predetermined end date for the data sharing.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Access Criteria: Data will be available for any research purpose to all interested parties who have approval from an independent review committee and who have a methodological sound proposal as determined by the steering committee of the current trial. Only the methodological qualities and not the purpose or objective of the proposal will be considered. Interested parties will be able to request the data by contacting the principal investigator. Authorship of publications emerging from the shared data will follow standard authorship guidelines from the International Committee of Medical Journal Editors and might or might not include authors from the steering committee depending on the nature of their involvement.